CLINICAL TRIAL: NCT05481424
Title: Light, Health, and Productivity: Evaluating the Potentials of Biodynamic Lighting for Home Office Workers
Brief Title: Evaluating the Potentials of Biodynamic Lighting for Home Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Korrus Inc. (Unknown)
Responsible Party: Principal Investigator, Nina Sharp, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00015724
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Performance; Sleep; Alertness
Keywords: Biodynamic Lighting; Sleep; Remote workers; Cognitive performance; light spectrum

STUDY DESIGN:
Intervention Model Description: Investigators will examine a series of participants (N=25), each of whom will participate in a five-week experiment. Each participant will have a screening visit at their home. The study will be conducted over five successive one-week periods with two cohorts of participants experiencing the same series of lighting interventions. All data collection will be performed during the working days (Monday - Friday) when participants are exposed to the lighting in their home offices.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodynamic Condition followed by an Active Placebo Condition. (Experimental): Each lighting condition will last for two weeks (Weeks 2-3 or 4-5), be limited to the 10 workdays, and be active for 8 hours per day. The order of conditions will be randomized.
  Interventions: Other: Biodynamic; Other: Active Placebo
- Active Placebo Condition followed by Biodynamic Condition (Experimental): Each lighting condition will last for two weeks (Weeks 2-3 or 4-5), be limited to the 10 workdays, and be active for 8 hours per day. The order of conditions will be randomized.
  Interventions: Other: Biodynamic; Other: Active Placebo

INTERVENTIONS:
Other: Biodynamic — This will be a nine-hour lighting scheme that includes three modes: morning, noon, and afternoon. It mimics natural lighting by providing blue-enriched bright lighting in the morning and yellowish dimmed lighting in the afternoon. The lighting scheme is designed to satisfy the visual lighting needs of office workers while maintaining a robust circadian clock.
Other: Active Placebo — We will include an active placebo condition that will be a whole-day lighting scheme with constant color and brightness during working hours. This condition is designed to serve to requirements: (1) to simulate a conventional, well-lit office lighting in compliance with the WELL standard V1 recommendations for circadian lighting design, and (2) to provide an Equivalent Melanopic Lux (EML) equal to the geometric average of EML delivered by the Biodynamic condition. Participants will receive a similar dose of lighting under both the Placebo and Biodynamic conditions; however, the "time" factor is ignored in the Placebo, and hence the method of delivery is different (constant versus dynamic).

SUMMARY:
This study examines the effectiveness of a biodynamic lighting intervention on the sleep, cognitive functions, and alertness of adults working from home. The biodynamic intervention is an innovative lighting solution that intends to harness both visual and non-visual effects of lighting through delivering varying intensities and spectra during working hours according to a preset protocol.

DETAILED DESCRIPTION:
The practice of working from home was widespread well before the 2020 Covid-19 pandemic; The Covid-19 pandemic pressed the fast-forward button on this trend. One of the biggest business concerns associated with working from home is how to maintain employees' productivity. Lighting has been proven as the main environmental element that significantly impacts office workers' health, sleep, mood, comfort, cognitive functions, and, consequently, productivity. One unintended aspect of working from home is the reduction in light exposure, especially in the contrast between the daytime and evening.

The effect of lighting on the office workers, including those working from home, could be roughly divided into two categories: visual route and non-visual route. Both visual and non-visual routes have received significant attention from researchers over the past decade. Yet, current literature lacks research involving a comprehensive approach that systematically evaluates the potential of biodynamic lighting interventions in home workplaces. None of the previous studies have evaluated lighting conditions in the home workplaces nor investigated the effects of lighting interventions on the health and productivity of adults working from home. With the rapid increase in the number of people moving to work from home, special attention should be paid to the lighting condition in home offices and its impacts on these workers.

This study examines the effectiveness of a biodynamic lighting intervention on the sleep, cognitive functions, and alertness of adults working from home. The biodynamic intervention is an innovative lighting solution that intends to harness both visual and non-visual effects of lighting through delivering varying intensities and spectra during working hours according to a preset protocol. Additionally, this study aims to compare the homeworkers' lighting conditions, impacts, and daily light exposure and how it is relevant to their sleep pattern and health. The specific aims of this study include:

* Aim 1: Examine the potential benefits of applying a biodynamic lighting condition in home offices for promoting sleep, cognitive functions, and alertness in remote workers.
* Aim 2: Objectively explore remote workers' daily light exposure pattern and model its relationship with their sleep quality.

Findings from this interdisciplinary study will provide insight into the potential benefits of applying biodynamic lighting in home workplaces for improving health and well-being in remote workers. Findings will also assist the lighting industry in providing necessary lighting technology and products aligned with the uprising trend of working from home.

ELIGIBILITY:
Inclusion Criteria:

* Have an occupation of a dayshift (i.e., occurring between 6 AM and 8 PM) remote office worker, working from home for five days (Monday→Friday) a week with a maximum of 12 hours per day
* Good health [self-reported medical history]
* No evidence of sleep disorders [Pittsburgh Sleep Quality Index (PSQI) scores >5 are excluded]
* No extreme chronotypes (extreme owl or lark) [Morningness-Evningness Questionnaire (MEQ) scores >70 or <30 are excluded; typical bedtime between 8 PM and 2 AM]
* Normal color vision [as per Ishihara's Tests for Colour Deficiency]
* No current or planned use of light therapy or light-altering devices (e.g., blue-blocking and/or tinted glasses and contact lenses)
* No planned upcoming travel during the study participation period
* Not pregnant

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Nocturnal Sleep Duration (in minutes) as measured by actigraphy | 24 hours everyday up to week 5
  Nocturnal Sleep Duration (in minutes) will be measured by Actigraphy. Longer sleep duration corresponds to improved sleep outcomes.
Change in Percent Sleep Efficiency (total sleep time divided by time in bed) measured by actigraphy | 24 hours everyday up to week 5
  Percent Sleep Efficiency measured by actigraphy. Higher percentage corresponds to higher sleep quality.
Change in the Subjective Sleep quality as measured by a single Likert-like question qualitatively | everyday up to 5 weeks
  This is included in the consensus sleep diary and consists of 1 question that is scaled from 1 to 7, with higher score corresponds to poor quality sleep.
Change in working memory as assessed by fractal 2-back score | Once per day, Monday to Friday, during week 1, 3, and 5
  Fractal 2-back score is based on number of correct responses. Higher test scores indicates better performance of working memory
Change in working Memory as assessed by Visual Object Learning Task (VOLT) score | Once per day, Monday to Friday, during week 1, 3, and 5
  Participants first memorize a set of 3-dimensional Euclidean shapes. During recall, participants are to distinguish between the initial shapes mixed with ten distractor shapes. Score is based on number of correct responses.
Change in median reaction time on Psychomotor Vigilance test | Once per day, Monday to Friday, during week 1, 3, and 5
  Psychomotor vigilance test(PVT) measures alertness and vigilant attention and is considered to be the gold standard measure of neurobehavioral effects of circadian misalignment and sleep loss. A shorter median reaction time corresponds to more attentive state.
Change in Balloon Analogue Risk Task (BART) score | Once per day, Monday to Friday, during week 1, 3, and 5
  Participants inflate balloons of unknown popping probability to obtain the highest reward. Each pump increases the potential reward. The potential reward is lost if the balloon pops. Scores are calculated by adding the number of pumps for unexploded balloons, with higher scores reflecting greater risk-taking. Range varies - explosions are at a random point between 1 and 128 pumps.
Change in subjective alertness as assessed by Stanford Sleepiness Scale (SSS) | Once per day, Monday to Friday, during week 1, 3, and 5
  SSS is a s self-reported Likert-type sleepiness scale which assess mental and physical sedation and sleepiness, respectively, at that moment and time. SSS only consists of 1 question that is scaled from 1 to 7, with 7 being a higher or worse score (i.e. more sleepy and sedated)

SECONDARY OUTCOMES:
Change in motor speed as assessed by Motor Praxis Task | Once per day, Monday to Friday, during week 1, 3, and 5
  Participants are to quickly touch ever-shrinking boxes. Each time a new box appears in a different location on the screen. A shorter reaction time corresponds to higher sensory motor speed.
Change in measure of abstraction: score on abstract matching test | Once per day, Monday to Friday, during week 1, 3, and 5
  Participants select pairs of shapes that fit with another shape. Higher number of correct responses corresponds to higher measure of abstraction.
Change in the spatial orientation: score on line orientation test | Once per day, Monday to Friday, during week 1, 3, and 5
  Participants are shown two lines at different angles, and are to rotate one line incrementally until it is parallel to the other. Higher scores corresponds to better spatial orientation.
Change in complex scanning and visual tracking: score on Digit Symbol Substitution Task (DSST) | Once per day, Monday to Friday, during week 1, 3, and 5
  Participants touch the number paired to the symbol that matches the current target symbol. Higher score corresponds to better complex scanning and visual tracking capability.

CONTACTS AND LOCATIONS:
Overall Officials: nina Sharp, PhD, Principal Investigator — Arizona State University
Locations (1):
- ASU DeSmart Lab, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. Results will be published by the investigators in academic journals and conference proceedings. However, neither the name nor identity of the participants will be used in any publications. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested in human-light interactions.
Time Frame: The data will be available after the data collection and analysis is complete which is anticipated to be in January 2024. The findings will be published in academic journals.